CLINICAL TRIAL: NCT05927610
Title: Evaluating the Role of Cerebrospinal Fluid (CSF) Cell-free DNA (cfDNA) as a Prognostic Biomarker in Glioblastoma
Brief Title: Genetic Testing of Cerebrospinal Fluid to Diagnose and Monitor Glioblastoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment has not yet been initiated
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-058
Record Dates: First submitted 2023-06-19; First posted 2023-07-03 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; CSF cfDNA; cerebrospinal fluid cell free DNA; Memorial Sloan Kettering Cancer Center; 23-058
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Cohort A will consist of newly diagnosed patients with Glioblastoma. Eligibility for enrollment prior to pathology diagnosis will be determined by a consensus diagnosis of high grade glioma based on clinical and radiographic evidence between neuroradiologist, neurosurgeon and study PI.
  Interventions: Diagnostic Test: Lumber Puncture
- Cohort B (Experimental): Cohort B will consist of patients with a histologically confirmed diagnosis of IDH WT glioblastoma.
  Interventions: Diagnostic Test: Lumber Puncture

INTERVENTIONS:
Diagnostic Test: Lumber Puncture — During the lumbar puncture/LP, 20cc will be collected per standard practice in adult patients. LP will be performed either at bedside or under interventional radiology (IR) guidance (due to patient anatomy).
  Other Names: LP

SUMMARY:
The goal of this study is to determine the utility of cerebrospinal fluid (CSF) cell-free DNA (cfDNA) as a prognostic biomarker in glioblastoma (GBM).

ELIGIBILITY:
Inclusion Criteria:

Cohort A

* Participants must be able to understand and be willing to sign a written informed consent document
* Age ≥ 18 years
* MRI with contrast-enhancing lesion concerning for high-grade glioma in absence of known systemic malignancy
* Clinical consensus of presumed diagnosis of high grade glioma between (1) neuroradiology (2) neurosurgery; and (3) principal investigator
* No prior tumor directed therapy
* Planned radiation therapy for glioblastoma
* Patients must be willing and able to tolerate MRI scans and/or CT scans w/ contrast
* Patients must be willing to consent to MSK IRB#12-245

Cohort B

* Participants must be able to understand and be willing to sign a written informed consent document
* Age ≥ 18 years
* Histologic confirmed glioblastoma (WHO grade IV), IDH wild type per IHC
* No prior tumor-directed therapies except surgical resection or biopsy
* Patients who have gliadel wafers placed during upfront surgery are excluded
* Planned radiation therapy for glioblastoma
* Patients must be willing and able to tolerate MRI scans and/or CT scans w/ contrast
* Patients must be willing to consent to MSK IRB#12-245

Exclusion Criteria:

Cohorts A and B

* Any case for which there is a medical contraindication or safety concern regarding a lumbar puncture under standard medical guidelines at MSK
* Refusal to undergo serial lumbar punctures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 6 months
  Overall survival will be calculated as the time from pathological diagnosis to the date of death due to any cause (prior to analysis cut-off) or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Miller, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org